CLINICAL TRIAL: NCT04222985
Title: Safety and Efficacy of 4 Investigational HSV 2 Vaccines Administered by Intramuscular Route in Adults With Recurrent Genital Herpes Caused by HSV 2
Brief Title: Safety and Efficacy of 4 Investigational HSV 2 Vaccines in Adults With Recurrent Genital Herpes Caused by HSV 2
Acronym: HSV15
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business reasons-Phase 2/Part B not conducted. Study terminated after last patient enrolled in Phase 1/Part A
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSV15; U1111-1183-6522 (Other: UTN)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (20):
- Part A - Group 1 (Experimental): HSV 2 formulation 1 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 1; Biological: Sodium Chloride 0.9%
- Part A - Group 2 (Experimental): HSV 2 formulation 2 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 2; Biological: Sodium Chloride 0.9%
- Part A - Group 3 (Experimental): HSV 2 Formulation 3 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 3; Biological: Sodium Chloride 0.9%
- Part A - Group 4 (Experimental): HSV 2 Formulation 4 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0, then HSV 2 Formulation 3 administered with concomitantly with 0.9% sodium chloride in the opposite arm at Month 2
  Interventions: Biological: HSV 2 Formulation 3; Biological: HSV 2 Formulation 4; Biological: Sodium Chloride 0.9%
- Part A - Group 5 (Experimental): HSV 2 Formulation 5 administered in one arm and Formulation 3 in the opposite arm, at Month 0 and Month 2.
  Interventions: Biological: HSV 2 Formulation 3; Biological: HSV 2 Formulation 5
- Part A - Group 6 (Placebo Comparator): Sodium chloride 0.9% (in both arms) at Month 0 and Month 2
  Interventions: Biological: Sodium Chloride 0.9%
- Part B (Stage 1) - Group 1 (Experimental): HSV 2 Formulation 1 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 1; Biological: Sodium Chloride 0.9%
- Part B (Stage 1) - Group 2 (Experimental): HSV 2 Formulation 2 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 2; Biological: Sodium Chloride 0.9%
- Part B (Stage 1) - Group 3 (Experimental): HSV 2 Formulation 3 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 3; Biological: Sodium Chloride 0.9%
- Part B (Stage 1) - Group 4 (Experimental): HSV 2 Formulation 4 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0, then HSV 2 Formulation 3 administered with concomitantly with 0.9% sodium chloride in the opposite arm at Month 2
  Interventions: Biological: HSV 2 Formulation 3; Biological: HSV 2 Formulation 4; Biological: Sodium Chloride 0.9%
- Part B (Stage 1) - Group 5 (Experimental): HSV 2 Formulation 5 administered in one arm and Formulation 3 in the opposite arm, at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 3; Biological: HSV 2 Formulation 5
- Part B (Stage 1) - Group 6 (Placebo Comparator): Sodium Chloride 0.9% (in both arms) at Month 0 and Month 2
  Interventions: Biological: Sodium Chloride 0.9%
- Part B (Stage 1) - Group 7 (Experimental): HSV 2 Formulation 6 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 6; Biological: Sodium Chloride 0.9%
- Part B (Stage 2) - Group 1 (Experimental): HSV 2 Formulation 1 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 1; Biological: Sodium Chloride 0.9%
- Part B (Stage 2) - Group 2 (Experimental): HSV 2 Formulation 2 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 2; Biological: Sodium Chloride 0.9%
- Part B (Stage 2) - Group 3 (Experimental): HSV 2 Formulation 3 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 3; Biological: Sodium Chloride 0.9%
- Part B (Stage 2) - Group 4 (Experimental): HSV 2 Formulation 4 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0, then HSV 2 Formulation 3 administered with concomitantly with 0.9% sodium chloride in the opposite arm at Month 2
  Interventions: Biological: HSV 2 Formulation 3; Biological: HSV 2 Formulation 4; Biological: Sodium Chloride 0.9%
- Part B (Stage 2) - Group 5 (Experimental): HSV 2 Formulation 5 administered in one arm and Formulation 3 in the opposite arm, at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 3; Biological: HSV 2 Formulation 5
- Part B (Stage 2) - Group 6 (Placebo Comparator): Sodium Chloride 0.9% (in both arms) at Month 0 and Month 2
  Interventions: Biological: Sodium Chloride 0.9%
- Part B (Stage 2) - Group 7 (Experimental): HSV 2 Formulation 6 administered concomitantly with 0.9% sodium chloride in the opposite arm at Month 0 and Month 2
  Interventions: Biological: HSV 2 Formulation 6; Biological: Sodium Chloride 0.9%

INTERVENTIONS:
Biological: HSV 2 Formulation 1 — Route of administration: Intramuscular
  Arms: Part A - Group 1; Part B (Stage 1) - Group 1; Part B (Stage 2) - Group 1
Biological: HSV 2 Formulation 2 — Route of administration: Intramuscular
  Arms: Part A - Group 2; Part B (Stage 1) - Group 2; Part B (Stage 2) - Group 2
Biological: HSV 2 Formulation 3 — Route of administration: Intramuscular
  Arms: Part A - Group 3; Part A - Group 4; Part A - Group 5; Part B (Stage 1) - Group 3; Part B (Stage 1) - Group 4; Part B (Stage 1) - Group 5; Part B (Stage 2) - Group 3; Part B (Stage 2) - Group 4; Part B (Stage 2) - Group 5
Biological: HSV 2 Formulation 4 — Route of administration: Intramuscular
  Arms: Part A - Group 4; Part B (Stage 1) - Group 4; Part B (Stage 2) - Group 4
Biological: HSV 2 Formulation 5 — Route of administration: Intramuscular
  Arms: Part A - Group 5; Part B (Stage 1) - Group 5; Part B (Stage 2) - Group 5
Biological: HSV 2 Formulation 6 — Route of administration: Intramuscular
  Arms: Part B (Stage 1) - Group 7; Part B (Stage 2) - Group 7
Biological: Sodium Chloride 0.9% — Route of administration: Intramuscular
  Arms: Part A - Group 1; Part A - Group 2; Part A - Group 3; Part A - Group 4; Part A - Group 6; Part B (Stage 1) - Group 1; Part B (Stage 1) - Group 2; Part B (Stage 1) - Group 3; Part B (Stage 1) - Group 4; Part B (Stage 1) - Group 6; Part B (Stage 1) - Group 7; Part B (Stage 2) - Group 1; Part B (Stage 2) - Group 2; Part B (Stage 2) - Group 3; Part B (Stage 2) - Group 4; Part B (Stage 2) - Group 6; Part B (Stage 2) - Group 7

SUMMARY:
The primary objectives of the study are:

* To describe the safety profile of different investigational vaccine regimens against herpes simplex virus type 2 (HSV-2).
* To evaluate the efficacy of the investigational vaccine regimens with respect to:
* the frequency of herpes simplex virus (HSV) deoxyribonucleic acid (DNA) detection in the genital area (shedding rate) following a 2 dose vaccine schedule
* the proportion of participants free of HSV genital recurrence at 6 months after the 2-dose vaccine schedule

The secondary objectives of the study are:

* To describe the impact of each of the investigational vaccine regimens in terms of total number of days with genital lesion up to 6 months after vaccination 2 and number of recurrences 60 days after the second vaccination compared with the placebo group
* To describe the efficacy of each of the investigational vaccine regimens with respect to the frequency of HSV DNA detection in the genital area (shedding rate) 60 days following the first vaccination visit plus 60 days following the second vaccination visit compared with the placebo group
* To describe the efficacy of each of the investigational vaccine regimens with respect to the frequency of HSV DNA detection in the genital area (shedding rate) 60 days following the first vaccination visit compared with the placebo group

DETAILED DESCRIPTION:
Study duration per participant is approximately 16 months

ELIGIBILITY:
Inclusion criteria :

* Aged 18 to 55 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* In good general health with absence of significant health problems as determined by medical history, physical examination, and laboratory screening performed during screening visits
* HSV-2 seropositive confirmed by Western blot
* A history of established HSV-2 infection ≥ 1 year
* A history of at least 2 and no more than 9 reported HSV clinical recurrences in the prior 12 months, or, if currently on suppressive therapy, history of at least 2 and no more than 9 reported clinical recurrences in the 12 months prior to initiation suppressive therapy
* For Part A and Part B, the participant is willing to refrain from using suppressive antiviral therapy starting 5 days before the first vaccination visit and up to 6 months after the second vaccination visit; and for Part B, throughout the 3, 60-day swabbing periods, and up to 6 months after the second vaccination visit
* For Part A and Part B, the participant is willing to refrain from using antiviral therapy to treat recurrences starting 5 days before V01 and up to 6 months after the second vaccination visit; and for Part B, throughout the 3, 60-day swabbing periods (i.e., up to 60 days after the second vaccination visit)

Exclusion criteria:

* For Part A, the participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 6 months after the last vaccination. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.
* For Part B, the participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence with her/his partner from at least 4 weeks before the enrollment visit until at least 6 months after the last vaccination. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.
* Participants whose female partners are pregnant at the time of enrollment or plan to become pregnant between study entry through 12 weeks (for Part A) and 6 months (for Part B) after the second vaccination visit.
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Receipt of any vaccine in the 4 weeks preceding the first study vaccination or planned receipt of any vaccine in the 4 weeks before and/or following any trial vaccination except for influenza vaccination, which may be received at a gap of at least 2 weeks before or 2 weeks after any study vaccination
* Current alcohol abuse or drug addiction
* Positive serologic test or polymerase chain reaction for human immunodeficiency virus type 1 infection
* Positive hepatitis B surface antigen
* Positive antibody for hepatitis C virusribonucleic acid and positive hepatitis C test
* Severe active infection or serious HSV-2 related medical conditions on the day of enrollment that, in the opinion of the Investigator, would prevent study completion
* Active genital herpes determined by the presence of outbreaks (genital lesions) at the time of enrollment. A prospective subject should not be included in the trial until 24 hours after the outbreak has resolved (the lesions have completely disappeared)
* Hemoglobin, white blood cell count with differential, platelet count, renal function tests (serum creatinine, blood urea nitrogen), liver function tests, creatine phosphokinase and C-reactive protein screening laboratory results that fall into the range of values that are Grade 2 or greater as per the study toxicity grading scale for this study. Also the range of values that are Grade 1 and are deemed clinically significant in the opinion of the Investigator (Grade 1 values deemed not clinically significant may be enrolled at the Investigator's discretion)
* Previous vaccination against HSV infection with either the trial vaccine or another vaccine against HSV
* History of HSV infection of the eye (e.g., herpes simplex interstitial keratitis or uveitis)
* History of eczema herpeticum
* History of herpes-associated erythema multiforme
* History of lesions caused by HSV on either arm
* History of any autoimmune disorder
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Thrombocytopenia or bleeding disorder, contraindicating IM vaccination based on Investigator's judgment
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Known allergy or intolerance to nickel
* Known allergy or intolerance to acyclovir or valacyclovir
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Chronic illness or other conditions that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to the Investigator's judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4 °F ([≥ 38 °C]).

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events | Within 4 hours (participants in Part A) or 30 minutes (participants in Part B) after vaccination
  Unsolicited systemic adverse events occurring immediately after vaccination
Number of participants with solicited injection site and systemic reactions | Within 7 days after vaccination
  Injection site reactions: injection site pain, erythema, and swelling. Systemic reactions: fever, headache, malaise, myalgia, arthralgia and chills
Number of participants with unsolicited adverse events | Within 30 days after vaccination
  An unsolicited adverse event is an event that does not fulfill the conditions prelisted in the Case Report Book in terms of diagnosis and/or onset post-vaccination
Number of participants with medically-attended adverse events (MAAEs) | From Day 0 to Month 14
  An MAAE is a new onset or a worsening of a condition that prompts the participant to seek unplanned medical advice at a physician's office or Emergency Department
Number of participants with adverse events of special interest (AESIs) | From Day 0 to Month 14
  AESIs are collected throughout the study
Number of participants with serious adverse events (SAEs) | From Screening to Month 14
  SAEs are collected throughout the study
Number of participants with out-of-range biological test results | From Day 8 to Day 30
  Out-of-range biological test results area assessed at Days 8 and 30 after each vaccination and 15 days prior to second vaccination in Part A and Days 8 and 30 after each vaccination in Part B
Viral genital shedding rate | 60 days before first vaccination and 60 days after the second vaccination
  Relative change in HSV DNA detection frequency between swabs collected before the first vaccination and those collected after the second vaccination visit
Genital HSV recurrence | 6 months following the second vaccination
  Proportion of participants free of genital HSV recurrence following the second vaccination

SECONDARY OUTCOMES:
Genital lesion rate | 6 months after the second vaccination
  Total number of days that the participants who receive investigational product or placebo report genital herpes lesions following the second vaccination
Genital HSV recurrence | 60 days following the second vaccination
  Number of recurrences of genital HSV following the second vaccination in participants who receive investigational product or placebo. Recurrence is defined as the appearance of genital and perineal lesions (i.e., shingles, blisters, ulcers) in a previously asymptomatic participant. Regarding 2 separate episodes of recurrences, recurrence is defined as the presentation of a new lesion (or lesions) after a 1-day-minimum (≥ 24 hours) lesion-free period
Viral genital shedding rate after the first and second vaccination | 60 days before first vaccination, and 60 days after the first vaccination, plus 60 days after the second vaccination
  Relative change in HSV DNA detection frequency between swabs collected before the first vaccination visit and those collected 60 days after the first vaccination visit plus after the second vaccination visit in participants who receive investigational product or placebo
Viral genital shedding rate after the first vaccination | 60 days before and 60 days after the first vaccination
  Relative change in HSV DNA detection frequency between swabs collected before the first vaccination visit and those collected 60 days after the first vaccination visit in participants who receive investigational product or placebo
Change in serum HSV 2-antibody levels | Before and 30 days after the first and second vaccinations and 6 months after the second vaccination
  Change between pre-vaccination and post-first and second vaccinations
Change in level of HSV 2-specific cellular immune responses | Before and 8 days after the first and second vaccination and 6 months after the second vaccination
  Change between pre-vaccination and post-first and second vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (4):
- United States (4):
  - Research Centers of America-Site Number:8400010, Hollywood, Florida
  - Brigham and Womens Hospital-Site Number:8400003, Boston, Massachusetts
  - M3 Wake Research Inc-Site Number:8400006, Raleigh, North Carolina
  - University of Washington Virology Research Clinic-Site Number:8400001, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org